CLINICAL TRIAL: NCT01993160
Title: 18F-FCH-PET/MR in Staging of High-Risk Prostate Cancer: A Multiparametric Approach
Brief Title: 18F-FCH (Fluorocholine)-PET/MR in Staging of High-Risk Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Prostate Cancer Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-FCH-PET/MR
Record Dates: First submitted 2013-10-25; First posted 2013-11-25 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Prostate Cancer
Keywords: Fluorocholine (FCH); Positron emission tomography (PET); Magnetic resonance imaging (MRI)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluorocholine; Injections; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-FCH PET MR (Experimental): Integrated whole body PET-MR or PET-CT and separate whole body MRI with use of 18F-FCH as the molecular probe
  Interventions: Drug: Fluorocholine (18F-FCH) Injection; Radiation: PET scan; Radiation: Whole body MRI

INTERVENTIONS:
Drug: Fluorocholine (18F-FCH) Injection — Before the PET-CT scan, the tracer (fluorocholine/FCH) will be injected into a vein in your arm just before the scan. This is the agent we are investigating in this study (not part of the standard procedure)
Radiation: PET scan — A whole body PET scan will be performed, integrated with either whole body low dose CT or whole body MRI
Radiation: Whole body MRI — A whole body MRI scan will be performed. This may be integrated with PET scan or performed separately.

SUMMARY:
This is a single centre, single arm feasibility study of 18FCH PET-MR imaging for staging patients with high risk prostate cancer.

Study Hypothesis:

FCH-PET/MR will enable more accurate staging of patients with high risk prostate cancer as compared to conventional imaging.

DETAILED DESCRIPTION:
Up to 60% of patients treated with radical prostatectomy or external beam radiotherapy for prostate cancer will have biochemical failure at 5 years. This may be due to several reasons, including presence of sub-clinical metastases at time of local therapy.

Currently, patients with high risk prostate cancer are staged by MRI of the prostate (to assess local extent of disease), CT of the abdomen(to detect spread to lymph nodes) and bone scan (to assess for spread to bones). However, these standard imaging exams do not always identify all sites of disease. Recent research has suggested that performing positron emission tomography (PET) scanning with a tracer called fluorocholine (FCH) improves identification of lymph node and bone metastases in prostate cancer, resulting in more accurate diagnosis.

The main goal of this study is to find out whether staging high risk prostate cancer patients with FCH PET-CT and MRI of the whole body will improve detection of primary tumors and metastases compared to current standard imaging exams. Improved staging of patients with prostate cancer may impact patient care as it will help to select more appropriate therapy.

In this study, participants will undergo either combined PET/MRI or PET-CT and MRI after standard evaluations. The accuracy of each staging approach (standard vs. PET and MRI) will be evaluated. In addition, we will incorporate novel methods for data interpretation by creating imaging maps combining data from PET and MRI (termed "Multiparametric maps"). The goal of this novel approach is to find out whether mapping 2 or more characteristics of a tumor at the same time will improve tumor detection and accuracy of diagnosis.

About 40 men from the Princess Margaret Hospital will take part in this study. The study should take about 2 years to complete enrollment and the results should be known within 36 months of completion of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologic diagnosis of carcinoma of prostate
* High risk disease: defined as Gleason ≥8, or T3 disease, or PSA >20ng/mL
* No prior therapy for prostate cancer (surgery, radiation therapy, hormone therapy, chemotherapy).
* Ability to provide written informed consent to participate in the study

Exclusion Criteria:

* Prior surgery or radiation therapy for prostate cancer
* Prior or ongoing hormone or other systemic therapy for prostate cancer
* Inability to lie supine for 90 minutes
* Any contraindication to MR as per Joint Department of Medical Imaging policies.
* Impaired kidney function with glomerular filtration rate < 30ml/min
* Previous anaphylactic reaction to gadolinium or other contraindications to MR.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of prostate cancer foci detected with FCH PET/MR compared to MR alone. | 2 years

SECONDARY OUTCOMES:
Detection rate of lymph node and distant metastases in patients with high risk prostate cancer as compared to conventional imaging strategies (CT abdomen and bone scintigraphy). | 2 years

OTHER OUTCOMES:
Overall accuracy of multiparametric mapping of choline metabolism with various MR parameters in staging of patients with high risk prostate cancer as compared to conventional imaging strategies. | 2 years
Relationship of choline kinase activity in the primary tumor (as expressed by FCH uptake) to presence of hypoxia and expression of GLUT-1 transporter proteins in pathology specimens. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ur Metser, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, University Health Network, 610 University Ave., Toronto, Ontario, Canada